CLINICAL TRIAL: NCT02649959
Title: An Open-Label Extension Study of CM-AT for the Treatment of Children With Autism With All Levels of Fecal Chymotrypsin
Brief Title: An Open Label Study of CM-AT for the Treatment of Children With Autism
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Curemark (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00104/Open Label-Autism
Record Dates: First submitted 2015-11-12; First posted 2016-01-08 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Autism
Keywords: Autism; A long-term extension study in a pediatric population of children with autism.
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): CM-AT
  Interventions: Drug: CM-AT

INTERVENTIONS:
Drug: CM-AT — Single unit does powder of active substance (CM-AT) administered 3 times per day

SUMMARY:
This is a Phase III, open label extension study evaluating the continued safety and efficacy of CM-AT in pediatric patients with autism with all levels of fecal chymotrypsin.

DETAILED DESCRIPTION:
Autism is clearly a significant cause of disability in the pediatric population. Treatment is based on the observation that many children with autism do not digest protein. CM-AT is a proprietary enzyme that is designed as a granulated powder taken three times daily.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 and 8 years, inclusive, at the time of signing informed consent/assent in Sponsor 00103 Study
* Completion of the Sponsor's 00103 Study who continue to meet eligibility requirements
* Currently in the 00102 open label study and continue to meet eligibility requirements
* Subjects who initially qualified for 00103 screening, who subsequently failed Baseline entrance criteria for randomization (@Visit 1) Baseline assessment of the ABC eligibility requirement who continue to meet eligibility requirements
* Up to 20 subjects 9-17 years of age who directly enroll into this study, who meet the current Diagnostic and Statistical Manual for Mental Disorders (DSM-IV-TR) diagnostic criteria for Autistic Disorder (AD), screened by the SCQ and confirmed by the ADI-R

Exclusion Criteria:

* Patient weighing < 13kg
* Allergy to porcine products
* Previous sensitization or allergy to trypsin, pancreatin, or pancrelipase
* History of severe head trauma, as defined by loss of consciousness or hospitalization, skull fracture or stroke.
* Seizure within the last year prior to enrollment, or the need for seizure medications either at present or in the past.
* Evidence or history of severe, moderate or uncontrolled systemic disease
* Ongoing dietary restriction for allergy or other reasons except nut allergies. Lactose free is allowable but not dairy free.
* Inability to ingest the study drug / non-compliance with dosing schedule.
* Inability to follow the prescribed dosing schedule.
* Use of any stimulant or non-stimulant medication or medications given for attention deficit hyperactivity disorder (ADHD) must be discontinued 5 days prior to the initial randomized study period.
* Subjects taking an selective serotonin reuptake inhibitor (SSRI) must be on a stable dose for a minimum of 30 days prior to entering the study.
* History of premature birth <35 weeks gestation.
* Prior history of stroke in utero or other in utero insult.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 405 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Aberrant Behavioral Checklist: Subscale of Irritability / Agitation (ABC-I) at fecal chymotrypsin (FCT) levels less than or equal to 12.6 | Change from Baseline to each post-baseline visit, through study completion Week 72.

SECONDARY OUTCOMES:
Aberrant Behavior Checklist: Subscale of Lethargy / Social Withdrawal (ABC-L) at fecal chymotrypsin (FCT) levels less than or equal to 12.6 | Change from Baseline to each post-baseline visit, through study completion Week 72.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Pearson, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Robert Hendren, DO, Principal Investigator — University of California, San Francisco
Locations (31):
- United States (31):
  - Southwest Autism Research & Resource Center (S.A.R.R.C.), Phoenix, Arizona
  - University of Arizona, Pediatrics Multidisciplinary Research Unit, Tucson, Arizona
  - Arkansas Children'S Hosp. Research Institute (A.C.H.R.I.), Little Rock, Arkansas
  - N.R.C. Research Institute, Orange, California
  - M.I.N.D. Institute (Univ.of California, Davis), Sacramento, California
  - University of California (U.C.S.F.), San Francisco, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Yale Child Study Center, New Haven, Connecticut
  - Segal Institute For Clinical Research, North Miami, Florida
  - Advent Health -Lake Mary Pediatrics, Orange City, Florida
  - A.P.G. Research, Orlando, Florida
  - Research Institute of Deaconess Clinic, Newburgh, Indiana
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - L.S.U. Health Sciences Center, Shreveport, Louisiana
  - Detroit Clinical Research Center, P.C., Bingham Farms, Michigan
  - Children'S Specialized Hospital, Egg Harbor, New Jersey
  - Children's Specialized Hospital, Toms River, New Jersey
  - Clinical Research Center of Nj, Voorhees Township, New Jersey
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Richmond Behavioral Associates, Staten Island, New York
  - Montefiore Med.Cneter, Autism & Obsessive Compulsive Spectrum Program, The Bronx, New York
  - Duke Center For Autism and Brain Development, Durham, North Carolina
  - Cleveland Clinic Autism Center, Cleveland, Ohio
  - Omega Medical Research, Warwick, Rhode Island
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - Vanderbilt Universtiy Med.Center-Treatment&Research Inst. For Asd, Nashville, Tennessee
  - University of Texas, Houston-Behavioral & Biomedical Sciences, Houston, Texas
  - Focus Center of Clinical Research, Clinton, Utah
  - University of Virginia, Dept. of Psychiatry and Neurobehavioral Sciences, Charlottesville, Virginia
  - Neuroscience, Inc, Herndon, Virginia
  - Carilion Clinic-Virginia Tech, Carilion School of Medicine, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McPheeters ML, Warren Z, Sathe N, Bruzek JL, Krishnaswami S, Jerome RN, Veenstra-Vanderweele J. A systematic review of medical treatments for children with autism spectrum disorders. Pediatrics. 2011 May;127(5):e1312-21. doi: 10.1542/peds.2011-0427. Epub 2011 Apr 4. PMID 21464191
- [Background] Autism and Developmental Disabilities Monitoring Network Surveillance Year 2008 Principal Investigators; Centers for Disease Control and Prevention. Prevalence of autism spectrum disorders--Autism and Developmental Disabilities Monitoring Network, 14 sites, United States, 2008. MMWR Surveill Summ. 2012 Mar 30;61(3):1-19. PMID 22456193
- [Background] Peacock G, Amendah D, Ouyang L, Grosse SD. Autism spectrum disorders and health care expenditures: the effects of co-occurring conditions. J Dev Behav Pediatr. 2012 Jan;33(1):2-8. doi: 10.1097/DBP.0b013e31823969de. PMID 22157409
- [Background] Ganz ML. The lifetime distribution of the incremental societal costs of autism. Arch Pediatr Adolesc Med. 2007 Apr;161(4):343-9. doi: 10.1001/archpedi.161.4.343. PMID 17404130
- [Background] McElhanon BO, McCracken C, Karpen S, Sharp WG. Gastrointestinal symptoms in autism spectrum disorder: a meta-analysis. Pediatrics. 2014 May;133(5):872-83. doi: 10.1542/peds.2013-3995. PMID 24777214
- [Background] Buie T, Campbell DB, Fuchs GJ 3rd, Furuta GT, Levy J, Vandewater J, Whitaker AH, Atkins D, Bauman ML, Beaudet AL, Carr EG, Gershon MD, Hyman SL, Jirapinyo P, Jyonouchi H, Kooros K, Kushak R, Levitt P, Levy SE, Lewis JD, Murray KF, Natowicz MR, Sabra A, Wershil BK, Weston SC, Zeltzer L, Winter H. Evaluation, diagnosis, and treatment of gastrointestinal disorders in individuals with ASDs: a consensus report. Pediatrics. 2010 Jan;125 Suppl 1:S1-18. doi: 10.1542/peds.2009-1878C. PMID 20048083
- [Background] Samsam M, Ahangari R, Naser SA. Pathophysiology of autism spectrum disorders: revisiting gastrointestinal involvement and immune imbalance. World J Gastroenterol. 2014 Aug 7;20(29):9942-51. doi: 10.3748/wjg.v20.i29.9942. PMID 25110424
- [Background] Elsabbagh M, Divan G, Koh YJ, Kim YS, Kauchali S, Marcin C, Montiel-Nava C, Patel V, Paula CS, Wang C, Yasamy MT, Fombonne E. Global prevalence of autism and other pervasive developmental disorders. Autism Res. 2012 Jun;5(3):160-79. doi: 10.1002/aur.239. Epub 2012 Apr 11. PMID 22495912
- [Background] Wasfy M, Oyofo B, Elgindy A, Churilla A. Comparison of preservation media for storage of stool samples. J Clin Microbiol. 1995 Aug;33(8):2176-8. doi: 10.1128/jcm.33.8.2176-2178.1995. PMID 7559972
- [Background] Cavallini G, Benini L, Brocco G, Riela A, Bovo P, Pederzoli P, Angelini G, Pelle C, Bertelli G, Scuro LA. The fecal chymotrypsin photometric assay in the evaluation of exocrine pancreatic capacity. Comparison with other direct and indirect pancreatic function tests. Pancreas. 1989;4(3):300-4. doi: 10.1097/00006676-198906000-00005. PMID 2734275
- [Background] Matthews DM. Intestinal absorption of amino acids and peptides. Proc Nutr Soc. 1972 Sep;31(2):171-7. doi: 10.1079/pns19720033. No abstract available. PMID 4563292
- [Background] Coutinho AM, Oliveira G, Morgadinho T, Fesel C, Macedo TR, Bento C, Marques C, Ataide A, Miguel T, Borges L, Vicente AM. Variants of the serotonin transporter gene (SLC6A4) significantly contribute to hyperserotonemia in autism. Mol Psychiatry. 2004 Mar;9(3):264-71. doi: 10.1038/sj.mp.4001409. PMID 15094787
- [Background] Naushad SM, Jain JM, Prasad CK, Naik U, Akella RR. Autistic children exhibit distinct plasma amino acid profile. Indian J Biochem Biophys. 2013 Oct;50(5):474-8. PMID 24772971
- [Background] Williams K, Wheeler DM, Silove N, Hazell P. Selective serotonin reuptake inhibitors (SSRIs) for autism spectrum disorders (ASD). Cochrane Database Syst Rev. 2010 Aug 4;(8):CD004677. doi: 10.1002/14651858.CD004677.pub2. PMID 20687077
- [Background] Tang G, Gudsnuk K, Kuo SH, Cotrina ML, Rosoklija G, Sosunov A, Sonders MS, Kanter E, Castagna C, Yamamoto A, Yue Z, Arancio O, Peterson BS, Champagne F, Dwork AJ, Goldman J, Sulzer D. Loss of mTOR-dependent macroautophagy causes autistic-like synaptic pruning deficits. Neuron. 2014 Sep 3;83(5):1131-43. doi: 10.1016/j.neuron.2014.07.040. Epub 2014 Aug 21. PMID 25155956
- [Background] Balasubramanian MN, Butterworth EA, Kilberg MS. Asparagine synthetase: regulation by cell stress and involvement in tumor biology. Am J Physiol Endocrinol Metab. 2013 Apr 15;304(8):E789-99. doi: 10.1152/ajpendo.00015.2013. Epub 2013 Feb 12. PMID 23403946
- [Background] Fairclough PD, Hegarty JE, Silk DB, Clark ML. Comparison of the absorption of two protein hydrolysates and their effects on water and electrolyte movements in the human jejunum. Gut. 1980 Oct;21(10):829-34. doi: 10.1136/gut.21.10.829. PMID 7192244
- [Background] Arnold GL, Hyman SL, Mooney RA, Kirby RS. Plasma amino acids profiles in children with autism: potential risk of nutritional deficiencies. J Autism Dev Disord. 2003 Aug;33(4):449-54. doi: 10.1023/a:1025071014191. PMID 12959424
- [Background] Munasinghe SA, Oliff C, Finn J, Wray JA. Digestive enzyme supplementation for autism spectrum disorders: a double-blind randomized controlled trial. J Autism Dev Disord. 2010 Sep;40(9):1131-8. doi: 10.1007/s10803-010-0974-2. PMID 20204691
- [Background] Schreck KA, Williams K, Smith AF. A comparison of eating behaviors between children with and without autism. J Autism Dev Disord. 2004 Aug;34(4):433-8. doi: 10.1023/b:jadd.0000037419.78531.86. PMID 15449518
- [Background] Bailey DB Jr, Raspa M, Olmsted M, Holiday DB. Co-occurring conditions associated with FMR1 gene variations: findings from a national parent survey. Am J Med Genet A. 2008 Aug 15;146A(16):2060-9. doi: 10.1002/ajmg.a.32439. PMID 18570292
- [Background] Lecavalier L. An evaluation of the Gilliam Autism Rating Scale. J Autism Dev Disord. 2005 Dec;35(6):795-805. doi: 10.1007/s10803-005-0025-6. PMID 16283084
- [Background] Marcus RN, Owen R, Kamen L, Manos G, McQuade RD, Carson WH, Aman MG. A placebo-controlled, fixed-dose study of aripiprazole in children and adolescents with irritability associated with autistic disorder. J Am Acad Child Adolesc Psychiatry. 2009 Nov;48(11):1110-1119. doi: 10.1097/CHI.0b013e3181b76658. PMID 19797985
- [Background] Yerys BE, Wallace GL, Sokoloff JL, Shook DA, James JD, Kenworthy L. Attention deficit/hyperactivity disorder symptoms moderate cognition and behavior in children with autism spectrum disorders. Autism Res. 2009 Dec;2(6):322-33. doi: 10.1002/aur.103. PMID 19998356
- [Background] Schreck KA, Williams K. Food preferences and factors influencing food selectivity for children with autism spectrum disorders. Res Dev Disabil. 2006 Jul-Aug;27(4):353-63. doi: 10.1016/j.ridd.2005.03.005. Epub 2005 Jul 25. PMID 16043324
- [Background] Borowitz D. Update on the evaluation of pancreatic exocrine status in cystic fibrosis. Curr Opin Pulm Med. 2005 Nov;11(6):524-7. doi: 10.1097/01.mcp.0000181474.08058.b3. PMID 16217179
- [Background] Penn AH, Hugli TE, Schmid-Schonbein GW. Pancreatic enzymes generate cytotoxic mediators in the intestine. Shock. 2007 Mar;27(3):296-304. doi: 10.1097/01.shk.0000235139.20775.7f. PMID 17304111
- [Derived] Pearson DA, Hendren RL, Heil MF, McIntyre WR, Raines SR. Pancreatic Replacement Therapy for Maladaptive Behaviors in Preschool Children With Autism Spectrum Disorder. JAMA Netw Open. 2023 Nov 1;6(11):e2344136. doi: 10.1001/jamanetworkopen.2023.44136. PMID 38032645